CLINICAL TRIAL: NCT06504537
Title: Comparative Effects of Theragun Percussion Therapy and Compression Therapy on Pain, Neck Range of Motion and Quality of Life in The Patients With Migraine
Brief Title: Comparative Effects of Theragun Percussion Therapy and Compression Therapy in The Patients With Migraine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/02100
Record Dates: First submitted 2024-06-11; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Migraine
Keywords: neck stiffness; headache; PNF; strteching; compression therapy
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the study would be single blinded as the assessor of the study would be kept blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A: THERAGUN PERCUSSION THERAPY AND ROUTINE PHYSICAL THERAPY (Experimental): Patients will receive Theragun Percussion Therapy for 25 minutes along with Routine Physical Therapy Treatment for 20 minutes
  Interventions: Other: THERAGUN PERCUSSION THERAPY
- GROUP B: COMPRESSION THERAPY AND ROUTINE PHYSICAL THERAPY (Experimental): Compression therapy will be administered to the patients by migraine relief gel cap for 25 minutes during migraine attacks along with Routine Physical Therapy Treatment for 20 minutes.
  Interventions: Other: COMPRESSION THERAPY

INTERVENTIONS:
Other: THERAGUN PERCUSSION THERAPY — In Group A, Patients will receive Theragun Percussion therapy along with routine Physical Therapy Treatment. The range of motion of lateral flexion and forward flexion will take by using a bubble inclinometer. Then the patient will place in a sitting position with the shoulder area exposed. Percussion therapy by using the Theragun device will give by a specific order. Treatment will start with the percussion head applied at the origin and insertion heads of the trapezius, Rhomboid and scalene muscle for 3-4 minutes each. Following this the percussive Theragun applicator will applied with circular strokes along the length of the muscle for 3 minutes. The pressure of application will adjust to the subject's tolerance.
  Arms: GROUP A: THERAGUN PERCUSSION THERAPY AND ROUTINE PHYSICAL THERAPY
Other: COMPRESSION THERAPY — In Group B, Compression therapy will be administered to the patients by migraine relief gel cap for 25 minutes during migraine attacks. The cap will store in a freezer (15-18°C). At the onset of the migraine attacks, patients wore the cap and used it. We will choose 25 minutes as the time for application of the gel cap based on the results of two published studies.(23) Headache severity will measured by Visual Analogue Scale and pain relief will measured on a similar scale. Analgesic treatment will not take within 25 minutes after the onset of cold therapy. If patients did not experience adequate relief from the headache, we will allow them to use analgesics 25 minutes after the onset of cold therapy. The routine physical treatment will be same as in group A.
  Arms: GROUP B: COMPRESSION THERAPY AND ROUTINE PHYSICAL THERAPY

SUMMARY:
The aim of this study is to compare the effects of Theragun Percussion therapy and Compression Therapy on pain, neck range of motion and quality of life in the patients with Migraine

DETAILED DESCRIPTION:
Migraine is a type of unilateral headache characterized by recurrent attacks of moderate to severe pulsating pain which common symptoms include increased sensitivity to light, noise, nausea and vomiting. Mechanical scalp compression is the most commonly used for temporary relief of migraine pain that originates from dilated blood vessels in the scalp. Many percussive therapy devices are used for relax and soothe sore muscles as Theragun helps in instant relief migraine pain.

It will be a Single blinded randomized clinical trial. Non-probability convenience sampling technique will be used to recruit 56 participants of 18 to 50 years of age from Riphah Rehabilitation Care Centre and Sir Ganga Ram Hospital, Lahore. The participants will be then randomly assigned into two equal groups through random number generation table. In Group A, Percussion Therapy will be applied by Theragun device for 25 minutes in each session along with Routine Physical Therapy Treatment for 20 minutes. In Group B, the Compression Therapy will be applied by migraine relief Gel Cap which works as Compression device for head for 25 minutes in each session along with Routine Physical Therapy Treatment for 20 minutes. The treatment will be given for 5 times per week for 6 weeks. Outcome measures for pre and post evaluation will be Visual Analogue Scale (VAS) for pain assessment, Migraine Screening Quality of life Questionnaire (MS-Q) for quality of life, Neck Disability Index (NDI) for neck disability, Bubble Inclinometer for neck range of motion. The data will be analyzed using SPSS version 24.

ELIGIBILITY:
Inclusion Criteria:

1. Both Genders
2. 18 to 65 years' old
3. Migraine without Aura
4. Headache with nausea or vomiting and light/sound sensitivity
5. Unilateral Headache from past 3 months at least once a week
6. ICHD-3 Criteria of migraine

Exclusion Criteria:

1. Congenital Condition of cervical spine
2. Inability of neck to perform flexion-rotation test
3. Meningitis, deep vein thrombosis
4. other-type of headache
5. Headache attributed to trauma or injury to neck

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
International Classification of Headache Disorders (ICHD-3) | 6 weeks
  Using ICHD-3 can aid first-visit patients by providing extended likely categories and removing the requirement for underlying cause disease remission before headache diagnosis. One of the ICHD-3 criteria for diagnosing migraines is
  * the quality of the pulsating pain.
  * Moderate to severe levels of pain
  * Made worse by day-to-day ordinary activities

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | 6 weeks
  The Neck Impairment Index is the most commonly used questionnaire to evaluate neck pain impairment (NDI) The NDI consists of ten questions: two ask about symptoms, the remaining question concerns concentration, and the other seven center on functional tasks. The 20-item test looks at four areas: activities of daily living, pain severity, emotion/cognition, and neck function. These categories show how a patient's neck pain condition affects their ability to operate both physically and emotionally
Migraine Screening Quality of Life Questionnaire (MS-Q) | 6 weeks
  The five-item migraine screen questionnaire, or MS-Q, was developed for use in research and clinical settings including occupational medicine and the general public as well as occupational medicine practitioners. The questionnaire is based on the diagnostic criteria for migraines published by the International Headache Society (IHS). This structured questionnaire consists of five items, each with a yes/no binary response option.
  For every "NO" response, a score of 0 is given, and for every "YES" response, a score of
  1. A cut-off point of ≥4 indicates a migraine case and a total score of 5 indicates this.
Visual Analogue Scale (VAS) | 6 weeks
  The VAS for attention was used to measure the participants' self-reported level of difficulty in maintaining focus. The participants were instructed to write a mark on the line that most accurately expressed their feelings regarding the challenge of paying attention.rating fron 0 to 10. 0 for no pain and 10 for worst pain.

OTHER OUTCOMES:
Bubble Inclinometer | 6 weeks
  Range of-motion is measured with a Bubble Inclinometer. Position the inclinometer near the joint that has to be measured; rotate the dial until the scale reaches zero; proceed to move the joint over its range; and finally, determine the distance traveled directly from the dial.

CONTACTS AND LOCATIONS:
Overall Officials: hira jabeen, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelly DP, Strauss AW. Inherited cardiomyopathies. N Engl J Med. 1994 Mar 31;330(13):913-9. doi: 10.1056/NEJM199403313301308. No abstract available. PMID 8114864
- [Background] Ferrari MD, Goadsby PJ, Burstein R, Kurth T, Ayata C, Charles A, Ashina M, van den Maagdenberg AMJM, Dodick DW. Migraine. Nat Rev Dis Primers. 2022 Jan 13;8(1):2. doi: 10.1038/s41572-021-00328-4. PMID 35027572
- [Background] Andreou AP, Edvinsson L. Mechanisms of migraine as a chronic evolutive condition. J Headache Pain. 2019 Dec 23;20(1):117. doi: 10.1186/s10194-019-1066-0. PMID 31870279
- [Background] Allen SM, Mookadam F, Cha SS, Freeman JA, Starling AJ, Mookadam M. Greater Occipital Nerve Block for Acute Treatment of Migraine Headache: A Large Retrospective Cohort Study. J Am Board Fam Med. 2018 Mar-Apr;31(2):211-218. doi: 10.3122/jabfm.2018.02.170188. PMID 29535237
- [Background] Wanderley D, Valenca MM, de Souza Costa Neto JJ, Martins JV, Raposo MCF, de Oliveira DA. Contract-relax technique compared to static stretching in treating migraine in women: A randomized pilot trial. J Bodyw Mov Ther. 2020 Apr;24(2):43-49. doi: 10.1016/j.jbmt.2019.05.023. Epub 2019 May 22. PMID 32507151
- [Background] Nasb M, Qun X, Ruckmal Withanage C, Lingfeng X, Hong C. Dry Cupping, Ischemic Compression, or Their Combination for the Treatment of Trigger Points: A Pilot Randomized Trial. J Altern Complement Med. 2020 Jan;26(1):44-50. doi: 10.1089/acm.2019.0231. Epub 2019 Oct 3. PMID 31580695